CLINICAL TRIAL: NCT04075123
Title: Respiratory Management Of Extremely Preterm Neonates: Evidence Generation And Implementation By Comparative Effectiveness Research (CER) Using Real World Data (RWD) From A Practice-Based Research Network (PBRN)
Brief Title: CPAP vs NIPPV: A COMPARATIVE EFFECTIVENESS RESEARCH
Status: Completed | Type: Observational
Sponsor: Canadian Neonatal Network (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Prakesh Shah, Director, Canadian Neonatal Network
Other Study IDs: 2019-01
Record Dates: First submitted 2019-08-27; First posted 2019-08-30 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Respiratory Insufficiency Syndrome of Newborn
Keywords: CPAP; NIPPV; INFANT, PREMATURE; RESPIRATORY MANAGEMENT; POST-ESTUBATION
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CPAP GROUP: Suggested PEEP range 5-10 cmH2O; Minimum required PEEP WILL BE 8 cm water (7 cm water if using bubble CPAP); Maximum allowable† PEEP: 12 cmH2O
  Interventions: Other: CPAP
- NIPPV GROUP: Suggested Ranges: PIP 12 to 24 cm water; PEEP 5 to 10 cm water; Rates 20-40 bpm; iTime 0.4-1.0 seconds; Minimum required settings on NIPPV: PEEP 8 cm water; Difference of pressure 6 cm water; Rate 20 bpm; Maximum allowable settings: PEEP 10 cm water; PIP 24 cm water; Rate 60 bpm

INTERVENTIONS:
Other: CPAP — The two NRS strategies being compared will be initiated at the time of first extubation (NRS support practices prior to initial intubation will be as per local unit guidelines and practices) and all subsequent extubations (if applicable) until 32 weeks PMA. For instance, a unit adopting post-extubation NCPAP strategy will initiate this mode following the initial and all subsequent extubations until 32 weeks PMA whereas centres adopting post-extubation NIPPV will initiate NIPPV following initial and all subsequent extubations until 32 weeks PMA.
  Other Names: NIPPV
  Groups: CPAP GROUP

SUMMARY:
Aim: Investigators aim is to conduct two complementary and concurrent CER projects using a pragmatic clinical trial design and registry-based RWD to identify the optimal respiratory management practices for extremely preterm neonates and reduce the risk of BPD and SNI.

Objectives: Two complementary objectives are proposed. Objective 1: To determine the efficacy and safety of "mandatory non-extubation" until 72 hours of postnatal age for preterm neonates born at 23 -25 weeks' GA who receive mechanical ventilation.

Objective 2: To determine whether optimal nasal continuous positive airway pressure post-extubation is as efficacious as nasal intermittent positive pressure ventilation in preterm neonates born at 23 -28 weeks' GA who have received mechanical ventilation.

DETAILED DESCRIPTION:
Background and Importance: Preterm neonates <29 weeks' gestational age (GA) have a 10% risk of mortality, 15% risk of severe neurological injury (SNI) and 45% risk of bronchopulmonary dysplasia (BPD). Both SNI and BPD are associated with significant long-term impairment. Various management approaches to prevent these complications are adopted without rigorous evaluation because conducting large-scale randomized trials can be challenging. One area consistently associated with SNI and BPD is respiratory management of these neonates which is also the area lacking evidence-informed approach. Comparative effectiveness research (CER) of different management strategies using Real World Data (RWD) is suggested as an alternative to generate Real World Evidence (RWE). Hypotheses Evaluating Treatment Effectiveness (HETE) studies are a form of CER where two or more practices are compared to evaluate presence or absence of anticipated effect using specific hypothesis. In this proposal, investigators will study two specific respiratory management practices for preterm neonates <29 weeks' GA using this design under the auspices of our practice based research network of the Canadian Preterm Birth Network (CPTBN) which has extensive routine data collection for this population.

Aim: Investigators aim to conduct two complementary and concurrent CER projects using a pragmatic clinical trial design and registry-based RWD to identify the optimal respiratory management practices for extremely preterm neonates and reduce the risk of BPD and SNI.

Objectives: Two complementary objectives are proposed. Objective 1: To determine the efficacy and safety of "mandatory non-extubation" until 72 hours of postnatal age for preterm neonates born at 23 -25 weeks' GA who receive mechanical ventilation.

Objective 2: To determine whether optimal nasal continuous positive airway pressure post-extubation is as efficacious as nasal intermittent positive pressure ventilation in preterm neonates born at 23 -28 weeks' GA who have received mechanical ventilation.

Methods:

Approach: These two CER projects will compare respiratory management approaches at the unit-level allowing investigators to study all eligible preterm neonates admitted to participating units. Twenty units in Canada have agreed to participate in each project, and The units have participated in the conception of the study, standardizing two-arms of the protocol and agreed on the project-specific data requirements.

Duration: The study will run over 4 years. Sample size: Considering superiority approach investigators will study 800 neonates for project 1 (α=0.05, β=0.2, baseline rate 35-40% and 30% relative risk reduction).

If there was a true difference in risk of failure of 1% in CPAP group (30% vs 29%), then 1816 patients were required to be 80% sure that the upper limit of a one-sided 97.5% confidence interval (or equivalently a 95% two-sided confidence interval) would exclude a difference in favour of the NIPPV group of more than 5% for neonates of 23 -28 weeks' GA for project 2. (modification in Nov 2021, uploaded later)

Analyses: In order to generate information necessary for causal inference in a pragmatic experimental design, investigators will conduct three-pronged sensitivity analyses: logistic regression, propensity-score based analyses and instrumental variable analyses to confirm or refute our hypotheses and improve generalizability of results. Expertise: The research team includes the expertise of clinicians, researchers, epidemiologists, knowledge users, parents and statisticians.

Expected outcomes: Through use of RWD collected by the CPTBN and HETE design, the proposal will result in identifying a superior respiratory management strategy and reduced risk of mortality, SNI, and BPD for extremely preterm neonates.

ELIGIBILITY:
Inclusion Criteria: Must meet all criteria

1. Preterm neonates <29 weeks gestational age
2. Receipt of mechanical ventilation

Exclusion Criteria:

1. Not received mechanical ventilation or active care
2. Congenital/genetic/chromosomal anomalies

Ages: 23 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates <29 weeks gestational age (including outborns) who have required mechanical ventilation at any time during their clinical course.
Sampling Method: Non-Probability Sample
Enrollment: 1829 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Failure on assigned NRS mode within 72 hours post-initial extubation | 72 hours
  * CPAP arm
    * Switch to any one of: NIPPV (including NIV-NAVA), or NIHFV
    * Escalation of CPAP PEEP >12 cmH2O
    * Intubation
  * NIPPV arm
    * Switch to any one of: NIHFV or NIV-NAVA (for centres that use unsynchronized NIPPV as their primary post-extubation mode)
    * Escalation of NIPPV beyond any one or more of the maximum allowable settings as described earlier
    * Switch to CPAP with PEEP > calculated MAP on NIPPV
    * Intubation

SECONDARY OUTCOMES:
Failure on assigned NRS mode within 7 days post-initial extubation | 7 days
Need for intubation within 72 hours and 7 days post-initial extubation | 72 hours and 7 days
Bronchopulmonary dysplasia (BPD) at 36 weeks' PMA | 36 weeks post mestrual age
Mortality before hospital discharge | through study completion, an average of 14 weeks
PMA when off positive pressure support | through study completion, an average of 14 weeks
Days of EMV (Post-initial extubation) | through study completion, an average of 14 weeks
Days of non-invasive respiratory support including high flow (Post-initial extubation) | through study completion, an average of 14 weeks
Days of any respiratory support (Post-initial extubation) | through study completion, an average of 14 weeks
Days of supplemental oxygen requirement (Post-initial extubation) | through study completion, an average of 14 weeks
Chronological age and post-menstrual age at time of full enteral feeds | through study completion, an average of 14 weeks
Air leak (Post-initial extubation) | through study completion, an average of 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prakesh Shah, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We do not have mechanisms to ask patients to allow data sharing.